CLINICAL TRIAL: NCT05303363
Title: Monitoring of Cerebral Blood Flow in Patients on Extracorporeal Membrane Oxygenation
Acronym: NOTICE
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, A.P.J. Vlaar, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W21_486 # 21.539
Record Dates: First submitted 2022-02-10; First posted 2022-03-31 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Cerebral Circulatory Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VV-ECMO: Critically ill patients with a suspected indication for VV-ECMO. ECMO will be provided according to local guidelines. In the Amsterdam UMC, location AMC, next to VV-ECMO, veno-arterial (VA-ECMO) is also provided. For this study, only patients on VV-ECMO will be included.
  Interventions: Device: VV-ECMO

INTERVENTIONS:
Device: VV-ECMO — VV-ECMO is indicated in case of severe respiratory failure refractory to other therapies. Indications for VV-ECMO include severe pneumonia, acute respiratory distress syndrome (ARDS) (a.o. due to COVID-19) or near-drowning. ECMO is considered a 'last resort' therapy, in which other maneuvers - such as prone positioning and neuromuscular blockage - have shown to be insufficient. Patients are generally receiving invasive mechanical ventilation and are almost always unconscious, since due to the severe respiratory failure, high doses of sedatives and neuromuscular blockage are often applied to prevent further ventilator-induced damage. After the decision for VV-ECMO is made, the patient is directly cannulated in the ICU or OR following standard protocols.

SUMMARY:
Venovenous extracorporeal membrane oxygenation (VV-ECMO) is a supportive therapy, indicated in case of severe, possibly reversible pulmonary failure, refractory to conventional therapies. Despite advances, morbidity and mortality remain high. Severe neurological complications can occur during ECMO, but their exact etiology is not well understood. It is hypothesized that fast correction of severe hypercapnia, a common indication for venovenous ECMO, may be detrimental for the brain. The supposed mechanism is that fast correction of hypercapnia may result in massive cerebral vasoconstriction and impaired cerebral blood flow (CBF). In this prospective, observational study the aim is to quantify change in CBF during routine initial correction of severe hypercapnia during VV-ECMO. Furthermore, the investigators will record any other hemodynamic changes during VV-ECMO. The hypothesis is that a larger decline in PaCO2 will result in a larger decline of CBF.

ELIGIBILITY:
Inclusion Criteria: in order to be eligible to participate in this study, a subject must meet all of the following criteria:

* High suspicion of an indication for VV-ECMO;
* Arterial line present to enable blood sampling;
* Older than 18 years.

Exclusion Criteria:

* Subjects will be excluded if the cerebral blood flow cannot be measured using the transcranial Doppler
* VA-ECMO or ECPR;
* No possibility for neuromonitoring measurements due to technical difficulties, e.g. post-craniotomy, unsuitable transcranial window;
* No possibility for neuromonitoring measurements due to circumstantial difficulties, e.g. ECPR;
* Contraindications for ECMO;
* ECMO is initiated in another center.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with a suspected indication for VV-ECMO. ECMO will be provided according to local guidelines. In the Amsterdam UMC, location AMC, next to VV-ECMO, veno-arterial (VA-ECMO) is also provided. For this study, only patients on VV-ECMO will be included.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Cerebral Blood Flow (CBF) velocity using Transcranial Doppler Ultrasound (cm/sec) | Before,during and after start of VV-ECMO,consisting of:starting 1 hour in advance of ECMO initiation, continuing until a maximum of 1 hour after the last change in SGF. 24 hours after ECMO initiation another measurement of 30 minutes will be performed.
  Change in CBF after correction of extracellular (arterial) pH during ECMO

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Vlaar, MD PhD MBA, Principal Investigator — Department of Intensive Care, Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC, Amsterdam-Zuidoost, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided